CLINICAL TRIAL: NCT01624532
Title: A Phase 2 Study to Assess Dose-Response, Efficacy (Immunogenicity) and the Safety of GC1109 Administered in Multi Intramuscular Doses to Healthy Subjects
Brief Title: A Study to Assess Dose-Response, Efficacy (Immunogenicity) and the Safety of GC1109
Acronym: GC1109
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GC1109_P2; GC1109 (Registry Identifier: Green Cross Croporation)
Record Dates: First submitted 2012-03-06; First posted 2012-06-20 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Anthrax
Keywords: Anthrax vaccine
MeSH Terms: conditions — Anthrax | interventions — Replication Protein A

STUDY DESIGN:
Intervention Model Description: Step 1 (Number of Arms: 4), Step 2 (Number of Arms: 2)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC1109 (Experimental): Step1: GC1109 0.3 mL or 0.5 mL or 0.1mL administered in Multi Intramuscular Doses (3 times) to Healthy Subjects
  Step2: GC1109 1.0 mL administered in Multi Intramuscular Doses (4 times) to Healthy Subjects
  Interventions: Biological: GC1109 or Placebo of GC1109
- Placebo of GC1109 (Placebo Comparator): Step1: Placebo of GC1109 0.5mL administered in Multi Intramuscular Doses (3 times) to Healthy Subjects
  Step2: Placebo of GC1109 1.0 mL administered in Multi Intramuscular Doses (4 times) to Healthy Subjects
  Interventions: Biological: GC1109 or Placebo of GC1109

INTERVENTIONS:
Biological: GC1109 or Placebo of GC1109 — Step1: Administer 0.3mL or 0.5mL or 0.1mL or placebo of GC1109 into the deltoid muscle three times every four weeks.
  Step2: Administer 1.0mL of GC1109 or placebo of GC1109 into the deltoid muscle three times every four weeks, and once after 24 weeks.
  Other Names: rPA or Placebo

SUMMARY:
The purpose of this study is to Assess Dose-Response, Efficacy (Immunogenicity) and the Safety of GC1109 Administered in Multi Intramuscular Doses to Healthy Subjects.

DETAILED DESCRIPTION:
1. Step 1

   Primary objective
   * Investigate the optimum volume of GC1109 to compare the subject ratio after seroconversion in each Anti-PA Ab by TNA at 4 weeks following infuse the drug 3 times with the immunogenicity of each treatment (GC1109 and placebo cohort) in healthy adults.
   * In healthy adults, three times the clinical dose of about four weeks, compare immunogenicity of each treatment group (GC1109 group and the placebo group) with subsects ratio who have been Seroconversion for Anti-PA Ab by TNA

   Secondary objective
   * Percentage of subjects after seroconversion in each anti-PA IgG level (by ELISA) at 4 weeks following infuse the drug 3 times in healthy adults
   * Check the Seroprotection antibody titer (survival rate : 50%) with passive immune (nonclinical tests) at 4 weeks following infuse the drug 3 times in healthy adults
   * Establish the Seroconversion rate from the percentage of subjects after seroconversion at 4 weeks following infuse the drug 3 times and seroprotection antibody titer in healthy adults
   * Compare the immunogenicity of each treatment with the GMT's assessment of Anti-PA Ab by TNA for 4 weeks following infuse the drug 3 times
   * Compare the immunogenicity of each treatment with the GMT's assessment of Anti-PA IgG by ELISA for 4 weeks following infuse the drug 3 times
   * Determine the safety of the each treatment cohort
2. Step 2

Primary objective

• Evaluate whether the Toxin Neutralization Antibody by TNA assay satisfy the NF50 standard or not at 4 weeks following infuse the optimal dose of GC1109 4 times in healthy adults.

Secondary objective

* Establish the safety of the GC1109 in healthy adults
* Establish the GMT of Toxin Neutralization Antibody by TNA assay after infusing the drug 4 times until 24 weeks in healthy adults
* Establish the GMT of Anti-PA IgG by ELISA after infusing the drug 4 times until 24 weeks in healthy adults

ELIGIBILITY:
Step1

Inclusion Criteria:

* Healthy 18 to 55 year-olds of either sex
* Body mass index above 18.5kg/m2 or below 30kg/m2 at the screening time
* A medical history without clinically significant congenital or chronic disease at the screening test before administrating the study drug within 28 days
* Agreement to avoid pregnancy or use contraceptive measure between 1 week prior to first dose and the 4 weeks following the final administration
* Female subjects of childbearing age, have negative serum β-HCG prior to infuse the study drug within 7 days and urine test at the every pre-vaccine
* Signed, informed voluntarily consents the clinical trials
* Willingness and agreement to comply with the constraints of the study protocol and ability to understand the study
* Willingness and ability to return for all follow-up visits and blood draws for the duration of the study
* Subjects who can have the study vaccine administered into the deltoid muscle and don't have the tattoo
* Agreement to stop drinking for 7days following the administration of the each study vaccine
* Agreement not to donate the blood for 24 hours following the administration of the each study vaccine

Exclusion Criteria:

* Prior history of, or known exposure to any form of B.anthracis or any anthrax immunization
* Employment in an industry involved in contact with ruminant animals, slaughterhose workers, handle the animal raw hides or raw wool, veterinary sciences involving ruminant animals, suspect exposure to any form of B. or anthrax immunization producer and developer.
* HIV positive or syphilis HAV, HBV, HCV positive or suspect
* Clinically significant out-of-range of laboratory tests at screening including : hypernatremia, hyponatremia, hypopotassemia, hyperchloremia, hypoproteinemia
* Prior history of, immunodeficiency or clinically active autoimmune disease
* Subjects with a history of Guillain-Barre syndrome
* Subjects with hemophilia or being treated with an anticoagulant who are at increased risk of serious bleeding during intramuscular injection
* History or evidence of metastatic malignancy tumor for internal organs, blood or flesh
* Medical significant hypersensitivity or idiosyncratic reaction related to any medical product including study drug or with a history of anaphylaxis
* Subjects who have had an acute fever exceeding a body temperature of 38.0℃ within 72 hours prior to the administration of the study vaccine, or who have had a symptom suspicious for acute febrile disease within 14 days prior to the administration of the study vaccine.
* Individuals who have received or intend to receive medication within 30 days of injection of the any experimental drug
* Donation of blood within 30 days prior to administrate the study drug
* Subjects who have received or are scheduled for the treatment with the following drug within 120 days (except for inhaled, nasal or topical corticosteroid)
* Subjects who have received or are scheduled for the treatment with the following drug within 120 days (except for inhaled, nasal or topical corticosteroid)

  * Systemic immunosuppressant therapy, radiotherapy, a high dose of steroid at the similar dose level
  * Blood-derived products including immunoglobulin
* Systemic immunosuppressant therapy, radiotherapy, a high dose of steroid at the similar dose level Blood-derived products including immunoglobulin
* Subjects who have received or are scheduled for the treatment with the following drug within the specified period
* Pre-injection of the IP within 30 days: oriental medicine
* Pre-injection of the IP within 7 days: ethical the counter drug (ETC), over the counter
* History or suspect of drug abuse (Amphetamine, barbiturates, cocaine, opioids, benzodiazepines etc)
* Subject without safety for the administration of vaccine, who in the investigator's opinion are unsuitable for the study or disturb the assessment of clinical trials

Step2

Inclusion Criteria:

* Healthy 19 to 65 year-olds of either sex
* A medical history without clinically significant congenital or chronic disease at the screening test before administrating the study drug within 28 days.
* For woman of childbearing age who have not undergone sterilization operation and woman who have not been more than 12 months after menopause, those who agree to avoid pregnancy or use appropriate contraceptive measure for the duration of the study from within one week prior to the first clinical drug administration. Man, who agree to avoid pregnancy or use contraceptive measure for the duration of the study
* Female subjects of childbearing age, have negative in pregnancy test at the screening visit
* Signed, informed voluntarily consents the clinical trials
* Subjects who can have the study drug administered into the deltoid muscle and don't have the tattoo
* Agreement not to donate the blood for the duration of the study

Exclusion Criteria:

* Prior history of, or known exposure to any form of B. anthracis or any anthrax immunization
* Employees in an industry involved in contact with ruminant animals(slaughterhouse workers, handle the animal raw hides or raw wool, veterinary sciences involving ruminant animals, suspect exposure to any form of B. or anthrax), immunization producer and developer.
* HIV positive or suspect
* HAV, HBV, HCV positive or suspect
* Prior history of, immunodeficiency or clinically active autoimmune disease
* Subjects with a history of Guillain-Barre syndrome
* Subjects with hemophilia or being treated with an anticoagulant who are at increased risk of serious bleeding during intramuscular injection
* History or evidence of metastatic malignancy tumor for internal organs, blood or flesh
* Medical significant hypersensitivity, idiosyncratic reaction related to any medical product included in study drug or with a history of anaphylaxis
* Subjects who have had an acute fever exceeding a body temperature of 38.0℃ within 72 hours prior to the administration of the study vaccine, or who have had a symptom suspicious for acute febrile disease within 14 days prior to the administration of the study drug.
* A person who has received a split vaccine, inactivated vaccine, or actived vaccine within four weeks prior to administration of a study drug
* Subjects who have received or are scheduled for the treatment with the following drug within 120 days (except for inhaled, nasal or topical corticosteroid)

  * Systemic immunosuppressant therapy, radiotherapy, a high dose of steroid at the similar dose level
  * Blood-derived products including immunoglobulin
* A person who has a history of drug abuse within 6 months prior to the administration of a study drug or suspected of taking drugs for fear of abuse through questionnaire and physical examination
* Pregnant women and lactating women
* A person whom the investigator determined unsuitable for the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Step 1) Investigate the optimum volume of GC1109 | at 4 weeks following infuse the drug 3 times
  Investigate the optimum volume of GC1109 to compare the subject ratio after seroconversion in each Anti-PA Ab by TNA at 4 weeks following infuse the drug 3 times with the immunogenicity of each treatment (GC1109 and placebo cohort) in healthy adults.
Step 2) Toxin Neutralization Antibody (by TNA assay) of GC1109 | at 4 weeks following infuse the drug 4 times
  Percentage of subjects with an 0.56 or higher NF50 by evaluating Toxin Neutralization Antibody (by TNA assay) at 4 weeks following infuse the optimal dose of GC1109 4 times in healthy adults.

SECONDARY OUTCOMES:
Step 1) Percentage of subjects after seroconversion | for 4 weeks following infuse the drug 3 times
  Percentage of subjects after seroconversion in each anti-PA IgG level (by ELISA) at 4 weeks following infuse the drug 3 times in healthy adults
Step 1) Check the Seroprotection antibody titer | for 4 weeks following infuse the drug 3 times
  Check the Seroprotection antibody titer with passive immune (nonclinical tests) at 4 weeks following infuse the drug 3 times in healthy adults
Step 1) Seroconversion rate | for 4 weeks following infuse the drug 3 times
  Establish the Seroconversion rate from the percentage of subjects after seroconversion at 4 weeks following infuse the drug 3 times and seroprotection antibody titer in healthy adults
Step 1) Compare the immunogenicity with GMT by TNA | for 4 weeks following infuse the drug 3 times
  Compare the immunogenicity of each treatment with the GMT's assessment of Anti-PA Ab by TNA for 4 weeks following infuse the drug 3 times
Step 1) Compare the immunogenicity with the GMT by ELISA | for 4 weeks following infuse the drug 3 times
  Compare the immunogenicity of each treatment with the GMT's assessment of Anti-PA IgG by ELISA for 4 weeks following infuse the drug 3 times
Step 1), Step 2) Adverse Events | By 24 weeks following infuse the drug 4 times
  Adverse events such as subjective and objective symptoms
Step 2) GMT of Toxin Neutralization Antibody by TNA assay | By 24 weeks following infuse the drug 4 times
  Establish the GMT of Toxin Neutralization Antibody by TNA assay after infusing the drug 4 times until 24 weeks in healthy adults
Step 2)GMT of Anti-PA IgG by ELISA | By 24 weeks following infuse the drug 4 times
  Establish the GMT of Anti-PA IgG by ELISA after infusing the drug 4 times until 24 weeks in healthy adults

CONTACTS AND LOCATIONS:
Overall Officials: Nam Joong Kim, M.D., Principal Investigator — Seoul National University Hospital; Seong Heon Wie, M.D., Principal Investigator — Saint Vincent's Hospital, Korea; Won Suk Choi, M.D., Principal Investigator — Korea University Asan Hospital; Eun Jung Lee, M.D., Principal Investigator — Soonchunhyang University Hospital; Jacob Lee, M.D., Principal Investigator — Hallym University Medical Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea